CLINICAL TRIAL: NCT03163264
Title: Testing the Efficacy of a Technology-assisted Intervention to Improve Weight Management of Obese Patients Within Patient Aligned Care Teams at the VA
Brief Title: The Peer Assisted Lifestyle Intervention
Acronym: PAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IIR 15-378; 01607 (Other Grant/Funding Number: Veterans Administration)
Record Dates: First submitted 2017-05-19; First posted 2017-05-23 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Overweight
Keywords: obesity; weight loss; weight gain; weight management; primary care; health coach
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Weight Gain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PAL Intervention (Experimental): Body mass index of =30kg/m2 OR Body mass index of =25 kg/m2 with an obesity associated co-morbidity
  Receiving Peer Assisted Lifestyle intervention (PAL tool, health coaching at baseline, follow-up health coaching calls, potential support of goals from primary care provider)
  Interventions: Behavioral: Peer Assisted Lifestyle
- Enhanced Usual Care (EUC) (Active Comparator): Body mass index of =30kg/m2 OR Body mass index of =25 kg/m2 with an obesity associated co-morbidity
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Peer Assisted Lifestyle — Patients will use PAL online tool accessing weight management and lifestyle behaviors, and will meet with a health coach regularly to establish SMART goals.
  Other Names: PAL arm
  Arms: PAL Intervention
Behavioral: Enhanced Usual Care — Patients will be given information on "healthy living messages" that were created by the VA, and given more information on specific messages they are interested in from the health coaches, but will not receive official coaching. These messages are the current standard of care at the VA for obesity counseling.
  Other Names: EUC arm
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The PAL intervention uses a new software tool delivered on tablets to facilitate 5As-based weight management counseling with a peer health coach and the VA PACT healthcare team to promote goal-setting, behavior change, and weight loss in the primary care (PC) setting. The PAL intervention also includes 10-12 health-coaching calls to the patient over 12 months.

As part of a cluster-randomized controlled study, the investigators will randomize 17 primary care providers at the Brooklyn VA to receive either the PAL Intervention or an Enhanced Usual Care control. The primary aim of the study is to explore differences in feasibility, acceptability, and intermediate, behavioral, and weight loss outcomes at 6 and 12 months of 520 patients recruited from the randomized primary care providers.

Objective:

1) Explore the feasibility and impact of this intervention on intermediate, behavioral, and weight loss outcomes at 6 and 12 months post-intervention when compared to enhanced usual care.

DETAILED DESCRIPTION:
Veterans shoulder a disproportionate burden of obesity and its co-morbidities, including diabetes, hypertension, and hyperlipidemia. Modest weight loss in obese patients through diet and exercise improves health and prevents chronic disease, but primary care providers (PCPs) often fail to adequately counsel patients about their weight due to lack of time and training. Thus, tools and brief interventions are needed to support providers' behavior change counseling. The VA currently offers the MOVE! program to treat overweight and obese patients, but only 9% of eligible patients attend. At the same time, Veterans on average see their PCPs 3.6 times per year, which supports the importance of developing primary care (PC)-based interventions. The United States Preventive Services Task force (USPSTF) recommends the use of the 5As framework (Assess, Advise, Agree, Assist, Arrange) for counseling patients about weight.

Interactive behavior change technologies utilizing expert system software programs are an innovative way to facilitate 5As counseling to promote behavior change in primary care. These programs perform computerized risk, lifestyle, and theory- based, behavioral assessment to provide computer-generated, tailored advice to patients. They also can provide information to healthcare teams. The MOVE!11 software is an expert system program for VA patients referred to MOVE!, but is not currently used in primary care by Patient-Aligned Care Teams (PACT).

Collaborative goal setting can be used to achieve behavior change in this intervention. This construct, a critical component of several behavior change theories and models and corresponding to "agree" in the 5As model, has been widely recommended for health promotion in primary care. The investigators' formative work (MIRB #01333) using key informant interviews with PACT teamlets and MOVE! staff and focus groups with Veterans demonstrated that goal setting is feasible and acceptable to patients and PACT teamlets and provided insight on barriers to goal setting, and ways to facilitate goal-setting conversations.

During the development phase of this project, the investigators developed a primary care-based intervention called MOVE! Toward Your Goals (MTG) to facilitate weight management within primary care and increase adoption of intensive VA programs such as MOVE!. The PAL intervention uses the MTG software tool (that the investigators developed) delivered on tablets to facilitate 5As-based weight management counseling with a health coach and healthcare team to promote goal-setting, behavior change, and weight loss in the primary care setting. The Veteran also receives follow up with 10-12 health coaching calls over 1 year.

As part of a clustered randomized control trial, the investigators will randomize 17 primary care providers to either Enhanced Usual Care or the PAL Intervention, recruiting 520 subjects.

STUDY OBJECTIVES

* Test the impact of the PAL intervention on weight change and behavioral/clinical outcomes
* Identify predictors of weight loss in Veterans participating in the intervention group related to goal setting processes and intervention components
* Determine the impact of the PAL intervention on obesity-related counseling practices and attitudes

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 (this age range represents MOVE! eligibility)
* BMI of 30kg/m2 or a BMI of 25kg/m2 with obesity-associated condition
* Under the care of PCP with at least 1 prior visit with the provider in the past 24 months
* Access to a telephone
* Able to travel to Brooklyn VA for in-person evaluations at baseline, 6, and 12 months

Exclusion Criteria:

* Non-Veterans
* A documented current history of active psychosis, active bipolar disorder, or other cognitive issues via ICD-10 codes
* Undergoing insulin-therapy for diabetes
* Self-reported inability to read at a 5th grade level due to literacy level or vision problems
* Has attended more than 4 MOVE! sessions in the past year
* Pregnancy
* PCP stating that Veteran should not participate

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie R. Jay, MD MS, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wittleder S, Smith S, Wang B, Beasley JM, Orstad SL, Sweat V, Squires A, Wong L, Fang Y, Doebrich P, Gutnick D, Tenner C, Sherman SE, Jay M. Peer-Assisted Lifestyle (PAL) intervention: a protocol of a cluster-randomised controlled trial of a health-coaching intervention delivered by veteran peers to improve obesity treatment in primary care. BMJ Open. 2021 Feb 26;11(2):e043013. doi: 10.1136/bmjopen-2020-043013. PMID 33637544
- [Derived] Wittleder S, Wong L, Ruan AM, Illenberger N, Nicholson A, Portelli D, Cansler R, Tenner CT, Sherman SE, Aguilar AD, Sweat V, Orstad SL, Vandyousefi S, Fronshtein M, Smith S, Dixon A, Goldstein MG, Raffa SD, Wylie-Rosett J, Jay M. Peer Coaching to Support Weight Management in Primary Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2529136. doi: 10.1001/jamanetworkopen.2025.29136. PMID 40892413

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomization performed at provider level. Patients recruited from provider panels randomized to each arm (PAL or EUC).
Groups:
- PAL Intervention: Patients: Body mass index of =30kg/m2 OR Body mass index of =25 kg/m2 with an obesity associated co-morbidity
  Receiving Peer Assisted Lifestyle intervention (PAL tool, health coaching at baseline, follow-up health coaching calls, potential support of goals from primary care provider)
  Peer Assisted Lifestyle: Patients will use PAL online tool accessing weight management and lifestyle behaviors, and will meet with a health coach regularly to establish SMART goals.
- Enhanced Usual Care (EUC): Patients: Body mass index of =30kg/m2 OR Body mass index of =25 kg/m2 with an obesity associated co-morbidity
  Enhanced Usual Care: Patients will be given information on "healthy living messages" that were created by the VA, and given more information on specific messages they are interested in from the health coaches, but will not receive official coaching. These messages are the current standard of care at the VA for obesity counseling.
- PAL Intervention: Providers: Providers at Brooklyn VA with panel size > 250, Received training on the overview of the 5As and the intervention components and practiced brief MI (using role playing) to support Veterans' weight management goals and address barriers to change
- Enhanced Usual Care (EUC): Providers: Providers at Brooklyn VA with panel size > 250
Period: Overall Study
Arm/Group | PAL Intervention: Patients | Enhanced Usual Care (EUC): Patients | PAL Intervention: Providers | Enhanced Usual Care (EUC): Providers
Started | 120 | 161 | 10 | 10
Completed | 90 | 136 | 6 | 8
Not Completed | 30 | 25 | 4 | 2
Not completed — Withdrawal by Subject | 13 | 3 | 4 | 2
Not completed — Lost to Follow-up | 17 | 20 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients of Randomized Providers. If patients changed providers (due to attrition), then they were analyzed in the groups they were originally assigned. NOTE: Baseline data for providers were not collected except for sex.
Groups:
- PAL Intervention: Providers: Providers at Brooklyn VA with panel size > 250
  Providers received training on the overview of the 5As and the intervention components and practiced brief MI (using role playing) to support Veterans' weight management goals and address barriers to change.
- Enhanced Usual Care (EUC): Providers: Providers at Brooklyn VA with panel size > 250
  Providers did not receive additional training.
- Total: Total of all reporting groups
Arm/Group | PAL Intervention: Patients | Enhanced Usual Care (EUC): Patients | PAL Intervention: Providers | Enhanced Usual Care (EUC): Providers | Total
Number analyzed (Participants) | 120 | 161 | 10 | 10 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline data for providers were not collected except for sex
  years
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 51.6 (11.3) | 49.9 (11.6) |  |  | 50.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 5 | 6 | 71
  Male | 89 | 132 | 5 | 4 | 230
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline data for providers were not collected except for sex
  Participants
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    American Indian or Alaska Native | 2 | 3 |  |  | 5
    Asian | 3 | 2 |  |  | 5
    Native Hawaiian or Other Pacific Islander | 0 | 1 |  |  | 1
    Black or African American | 63 | 97 |  |  | 160
    White | 28 | 36 |  |  | 64
    More than one race | 6 | 5 |  |  | 11
    Unknown or Not Reported | 18 | 17 |  |  | 35
Region of Enrollment [Number; unit: participants] — Population: Baseline data for providers were not collected except for sex
  participants
    United States: number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    United States | 120 | 161 |  |  | 281
Height [Mean (Standard Deviation); unit: centimeters] — Population: Baseline data for providers were not collected except for sex
  centimeters
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 171.5 (8.9) | 173.8 (8.5) |  |  | 172.8 (8.8)
Weight [Mean (Standard Deviation); unit: kg] — Population: Baseline data for providers were not collected except for sex
  kg
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 98.9 (20.4) | 100.8 (16.3) |  |  | 100.0 (18.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Baseline data for providers were not collected except for sex
  kg/m^2
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 33.5 (5.6) | 33.3 (4.7) |  |  | 33.4 (5.1)
Waist Circumference [Mean (Standard Deviation); unit: inches (in)] — Population: Baseline data for providers were not collected except for sex
  inches (in)
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 42.9 (6.2) | 42.7 (4.7) |  |  | 42.8 (5.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Baseline data for providers were not collected except for sex.
  mmHg
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 79.3 (28.0) | 77.8 (10.5) |  |  | 78.5 (19.9)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Baseline data for providers were not collected except for sex
  mmHg
    number analyzed (Participants) | 120 | 161 | 0 | 0 | 281
    (all) | 123.8 (14.4) | 126.9 (41.9) |  |  | 125.6 (33.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight Change in Kg
Description: Weight change in kg at 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Groups:
- PAL Intervention: Body mass index of =30kg/m2 OR Body mass index of =25 kg/m2 with an obesity associated co-morbidity
  Receiving Peer Assisted Lifestyle intervention (PAL tool, health coaching at baseline, follow-up health coaching calls, potential support of goals from primary care provider)
  Peer Assisted Lifestyle: Patients will use PAL online tool accessing weight management and lifestyle behaviors, and will meet with a health coach regularly to establish SMART goals.
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
kilograms (kg) | -2.51 (0.73) | -0.79 (0.48)
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.050, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance. "Note: Estimated p-value was calculated at 0.050"; This analysis was in our grant and protocol paper but was added late to clinicaltrials.gov; Mean Difference (Net) = 0.05, 95% CI 2-sided [0 to 3.45]
Statistical Analysis 2: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney) — Statistical test was 2 sided with p<0.05 indicating statistical significance. "Note: Estimated p-value was calculated at 0.05"; The investigators will also use repeated measures modeling based on mixed models using baseline and follow up data to adjust for characteristics; Mean Difference (Net) = 0.05

2. Primary Outcome: Mean Percent Weight Change From Baseline to 12 Months
Description: Mann-Whitney tests for continuous outcomes (e.g., weight change)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
percent change | -2.32 (0.75) | -0.69 (0.47)
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.069, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; This analysis was in our grant and protocol paper but was added late to clinicaltrials.gov; Mean Difference (Net) = 0.069, 95% CI 2-sided [-0.13 to 3.39]
Statistical Analysis 2: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.028, Wilcoxon (Mann-Whitney) — Statistical test was 2 sided with p<0.05 indicating statistical significance; [statistical method as in outcome 1, analysis 2]; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [0.21 to 3.76]

3. Secondary Outcome: Achievement of 5% Weight Loss
Description: Percent of people in each arm attaining > or = to 5% weight loss
Time Frame: 6 months
Measure: Number; unit: Percent of people
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
Percent of people | 17 | 6
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.033, Mixed Models Analysis; Percent Difference = 11.18, 95% CI 2-sided [0.92 to 21.45]

4. Secondary Outcome: Achievement of 5% Weight Loss
Description: Percent of people in each arm attaining > or = to 5% weight loss
Time Frame: 12 months
Measure: Number; unit: Percent of people
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
Percent of people | 26 | 15
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.073, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Percent Difference = 11.08, 95% CI 2-sided [-1.05 to 23.2] — Adjusted

5. Secondary Outcome: Changes in HB A1C
Description: The investigators will extract HB A1C data from the electronic health record. Due to COVID, participants did not have their regular in-person doctor's appointments to test/collect their HB A1C. Due to a large amount of missing HB A1C data, data was not collected/extracted from the electronic health record and therefore changed in HB A1C was not analyzed.
Time Frame: 6 and 12 months
Population: Data were not collected.
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Changes in Waist Circumference
Description: To determine whether patients had changes in waist circumference. Adjusted changes between baseline and 6 Months. Mean (SD) of adjusted outcomes in each treatment arm are provided.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: inches (in)
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
inches (in) | -1.44 (0.31) | -0.72 (0.23)
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.065, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Mean Difference (Final Values) = 0.72, 95% CI 2-sided [-0.05 to 1.48]

7. Secondary Outcome: Changes in Waist Circumference
Description: To determine whether patients had changes in waist circumference. Adjusted changes between baseline and 12 Months. Mean (SD) of adjusted outcomes in each treatment arm are provided.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: inches (in)
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
inches (in) | -1.82 (0.37) | -1.40 (0.29)
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.378, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [-0.52 to 1.37]

8. Secondary Outcome: Changes in Physical Activity
Description: Measure duration and intensity using accelerometers. The ActiGraph Link (GT9X) accelerometer, worn on the wrist, was used to objectively measure PA for 7 days at Baseline, and at 6 and 12 months.
Time Frame: 6 and 12 months
Population: The investigators planned to use accelerometers, given out at each study visit, to measure physical activity for 7 days at baseline, 6 month, and 12 months. However, due to COVID-19, the investigators were unable to give out accelerometers at each visit to collect this data. Therefore, data collection was not completed and outcome will not be reported.
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Moderate to Vigorous Physical Activity Difference (Minutes)
Description: Measure duration using the Paffenbarger questionnaire items. Difference in adjusted mean behavioral outcome between the treatment arms. Adjusted mean difference (95% Confidence Interval) [p-value] between the treatment arms (PAL - EUC) for each behavioral outcome at 6 months of follow-up.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
minutes | 93.43 (57.88) | 101.78 (43.96)
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.911, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Mean Difference (Final Values) = 8.35, 95% CI 2-sided [-138.25 to 154.95]

10. Secondary Outcome: Moderate to Vigorous Physical Activity Difference (Minutes)
Description: Measure duration using the Paffenbarger questionnaire items. Difference in adjusted mean behavioral outcome between the treatment arms. Adjusted mean difference (95% Confidence Interval) [p-value] between the treatment arms (PAL - EUC) for each behavioral outcome at 12 (primary) months of follow-up.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
minutes | 13.32 (53.77) | 46.15 (45.34)
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.648, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Mean Difference (Final Values) = 32.83, 95% CI 2-sided [-108.15 to 173.81]

11. Secondary Outcome: Percent of People Achieving >150 Minutes of Vigorous to Moderate Physical Activity/Week
Description: Adjusted mean percent of people achieving behavioral outcome in each treatment arms. Measured duration using IPAQ questionnaire items.
Time Frame: 6 months
Measure: Number; unit: percent of people
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
percent of people | 70 | 80
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.736, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Percent Difference = 10.32, 95% CI 2-sided [-49.73 to 70.37]

12. Secondary Outcome: Percent of People Achieving >150 Minutes of Vigorous to Moderate Physical Activity/Week
Description: as for outcome 11
Time Frame: 12 months
Measure: Number; unit: percent of people
Arm/Group | PAL Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 120 | 161
percent of people | 29 | 49
Statistical Analysis 1: Comparison: PAL Intervention vs Enhanced Usual Care (EUC); Test type: Superiority; p = 0.53, Mixed Models Analysis — Statistical test was 2 sided with p<0.05 indicating statistical significance; Percent Difference = 19.36, 95% CI 2-sided [-41.09 to 79.8]

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were not monitored for providers.
Arm/Group | PAL Intervention: Patients | Enhanced Usual Care (EUC): Patients | PAL Intervention: Providers | Enhanced Usual Care (EUC): Providers
All-Cause Mortality (participants affected / at risk) | 0/120 | 2/161 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 14/120 | 17/161 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 36/120 | 51/161 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PAL Intervention: Patients (N=120) | Enhanced Usual Care (EUC): Patients (N=161) | PAL Intervention: Providers (N=0) | Enhanced Usual Care (EUC): Providers (N=0)
Shin bone fracture (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA — Shin bone fracture
Chest pain (Cardiac disorders) | 0 | 1 | NA | NA
Swollen nose (Infections and infestations) | 0 | 1 | NA | NA
Intestine infection (Infections and infestations) | 0 | 1 | NA | NA
Broken toe (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Broke vertebrae in neck (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Fainted (Metabolism and nutrition disorders) | 0 | 2 | NA | NA
Hernia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Stroke (Nervous system disorders) | 1 | 1 | NA | NA
Hip surgery (Surgical and medical procedures) | 0 | 1 | NA | NA
Feeding tube (Surgical and medical procedures) | 0 | 1 | NA | NA
Hernia surgery (Surgical and medical procedures) | 1 | 1 | NA | NA
Gall bladder removal (Surgical and medical procedures) | 0 | 1 | NA | NA
Back surgery (Surgical and medical procedures) | 0 | 1 | NA | NA
Infection (Infections and infestations) | 1 | 0 | NA | NA
Wrist pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Mental health check (Psychiatric disorders) | 1 | 0 | NA | NA
Respiratory issue (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Blood clot in lungs (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA | NA
Knee replacement (Surgical and medical procedures) | 1 | 0 | NA | NA
Fibroid removal (Surgical and medical procedures) | 1 | 0 | NA | NA
Prostate surgery (Surgical and medical procedures) | 1 | 0 | NA | NA
Surgery (Surgical and medical procedures) | 1 | 0 | NA | NA
Shoulder surgery (Surgical and medical procedures) | 1 | 1 | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PAL Intervention: Patients (N=120) | Enhanced Usual Care (EUC): Patients (N=161) | PAL Intervention: Providers (N=0) | Enhanced Usual Care (EUC): Providers (N=0)
Chest pain (Cardiac disorders) | 0 | 3 | NA | NA
Ear infection (Ear and labyrinth disorders) | 0 | 1 | NA | NA
Upset stomach (Gastrointestinal disorders) | 0 | 1 | NA | NA
Couldn't swallow (Gastrointestinal disorders) | 0 | 1 | NA | NA
Not feeling well (General disorders) | 1 | 1 | NA | NA
Allergic reaction (Immune system disorders) | 1 | 1 | NA | NA
Flu (Infections and infestations) | 2 | 2 | NA | NA
Tonsillitis (Infections and infestations) | 1 | 1 | NA | NA
Sore throat (Infections and infestations) | 0 | 1 | NA | NA
Head infection (Infections and infestations) | 0 | 1 | NA | NA
Bronchitis (Infections and infestations) | 0 | 2 | NA | NA
Infection (Infections and infestations) | 0 | 1 | NA | NA
Ankle sprain (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Work-related injury (Injury, poisoning and procedural complications) | 1 | 1 | NA | NA
Motor vehicle accident (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Sprained wrist (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Cut on finger (Injury, poisoning and procedural complications) | 2 | 1 | NA | NA
Dog bite (Injury, poisoning and procedural complications) | 0 | 1 | NA | NA
Diabetes (blurred vision/high sugar) (Metabolism and nutrition disorders) | 0 | 1 | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | NA | NA
Hand dysfunction (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Hernia (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Knee issue (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Knee, groin pull, back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Pain and couldn't walk (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Sciatica pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Arm pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Right shoulder tear (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Gout (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA | NA
Pain in sides (Musculoskeletal and connective tissue disorders) | 0 | 1 | NA | NA
Migraine (Nervous system disorders) | 1 | 1 | NA | NA
Depression (Psychiatric disorders) | 0 | 1 | NA | NA
Kidney pain/stones (Renal and urinary disorders) | 0 | 2 | NA | NA
Blood in urine and pain (Renal and urinary disorders) | 0 | 1 | NA | NA
Breathing issues (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | NA | NA
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | NA | NA
Elevated blood pressure (Vascular disorders) | 2 | 2 | NA | NA
High pulse and temperature (Cardiac disorders) | 1 | 0 | NA | NA
Blood vessel in eye (Eye disorders) | 1 | 0 | NA | NA
ED visit for medication (General disorders) | 1 | 0 | NA | NA
Tendinitis (Infections and infestations) | 1 | 0 | NA | NA
Laryngitis (Infections and infestations) | 1 | 0 | NA | NA
Excessive bleeding (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Eye injury (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Hand injury (Injury, poisoning and procedural complications) | 1 | 0 | NA | NA
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Neck issue (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA | NA
Headaches (Nervous system disorders) | 3 | 0 | NA | NA
Vertigo (Nervous system disorders) | 1 | 0 | NA | NA
Eating disorder (Psychiatric disorders) | 1 | 0 | NA | NA
Urinary tract infection (Renal and urinary disorders) | 1 | 0 | NA | NA
Skin issue (Skin and subcutaneous tissue disorders) | 1 | 0 | NA | NA

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic was a limitation that impacted recruitment and decreased our power to see significant differences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT03163264/Prot_SAP_000.pdf